CLINICAL TRIAL: NCT00992576
Title: A Confirmatory, Placebo-controlled, Randomised, Double-blind, Single-dummy, Parallel Group, Ratio-finding Study in Constipated Pain Patients to Establish an Optimal Hydromorphone - Naloxone Ratio With an Improved Bowel Function and a Comparable Analgesic Efficacy Compared to Hydromorphone Alone
Brief Title: Optimisation of Hydromorphone - Naloxone Ratio for the Treatment of Pain
Acronym: HMX3501
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-005312-18
Record Dates: First submitted 2009-10-06; First posted 2009-10-09 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Constipation
Keywords: Confirmatory; Constipation; Pain; Hydromorphone; Naloxone
MeSH Terms: conditions — Constipation; Pain

INTERVENTIONS:
Drug: Active Hydromorphone PR + Active Naloxone PR — Optimal pain relief and improved bowel function in constipated pain patients
Drug: Active Hydromorphone PR + Placebo Naloxone PR — Optimal pain relief and improved bowel function in constipated pain patients

SUMMARY:
The purpose of this study is to establish an optimal hydromorphone - naloxone ratio with an improved bowel function for constipated pain patients.

DETAILED DESCRIPTION:
Subjects suffering from cancer or non-cancer pain suffering from constipation cased or aggravated by opioids will be randomised to one of four ratios of hydromorphone PR plus naloxone PR or Hydromorphone PR plus placebo to investigate whether a hydromorphone/naloxone combination will lead to comparable analgesia, with a decrease in constipation, and to investigate the optimal dose ratio of hydromorphone and naloxone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years with a history of non-cancer or cancer pain that requires around-the-clock opioid therapy (8, 24 or 48 mg hydromorphone PR per day for the duration of the study).
2. Subjects with constipation caused or aggravated by opioids
3. Subjects must be willing to discontinue their current opioid analgesic routine, and .
4. current laxative regimen

Exclusion Criteria:

1. Chronic or intermittent pain that results from Fibromyalgia or Rheumatoid Arthritis.
2. Subjects presently taking, or who have taken, naloxone <=30 days prior to the start of the Screening Period.
3. Subjects suffering from diarrhoea.
4. Abnormal liver or kidney function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Bowel Function Measure Average pain scores

SECONDARY OUTCOMES:
Bowel Function Measures Rescue medication use

CONTACTS AND LOCATIONS:
Locations (14):
- Hunter New England Area Health Service, Newcastle, New South Wales, Australia
- AKH Wien - Universitätskliniken, Vienna, Austria
- Erasme Hospital, Brussels, Belgium
- Poradna pro lecbu bolesti, Příbram, Czechia
- Speciallæge Michael Crawford, København K., Denmark
- Oma Lääkäri Oy, Kuopio, Finland
- CHU - Hôpital Amiens Nord, Amiens, France
- Universitaetsklinikum Jena, Jena, Germany
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel
- Diakonessenhuis, locatie Zeist, Zeist, Netherlands
- Szpital Uniwersytecki w Krakowie Zakład Badania, Krakow, Poland
- Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca, Romania
- Kantonsspital Aarau, Aarau, Switzerland
- Avondale Surgery, Chesterfield, United Kingdom